CLINICAL TRIAL: NCT00345449
Title: Evaluation of a Decision Aid for Adult Cystic Fibrosis Patients Considering Bilateral Lung Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2004776-01
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis,; lung disease,; lung transplantation,; decision aid
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases | interventions — Decision Support Techniques

INTERVENTIONS:
Behavioral: Decision Aid

SUMMARY:
In 2006, the International Patient Decision Aids Collaboration (IPDAS) reached agreement on criteria for evaluation. Accordingly, the primary outcome is 'decision quality' 3 weeks after using the decision aid. Decision quality is defined as the extent to which a patient decision aid improves the match between the chosen option and the features that matter most to the informed patient. Measures include: a) patients' knowledge of essential facts [options, benefits, harms, and outcome probabilities]; and b. the congruence between the option chosen and patients' informed values regarding benefits and risks.

In the past twenty years lung transplantation has become the most widely accepted option of treating cystic fibrosis patients with severe lung disease. Lung transplantation can be a good experience for many patients, improving their quality of life and their survival. However there are potential risks of lung transplantation including infection, organ rejection and early death. Cystic fibrosis patients are often faced with making a choice of whether to be referred for lung transplantation when they are very sick and there is the immediate need to survive. Our group has developed a tool called a decision aid which we hope will assist the patient and family in making this choice. The decision aid guides the patient through a series of steps where they weigh the benefits and risks of being referred for lung transplantation and the benefits and risks of receiving 'usual care' without the option of referral.

DETAILED DESCRIPTION:
Patients randomized to either arm of the study will be required to undergo a lung transplantation education and counselling session with their CF physician prior to randomization. Subsequent to this session patients will be randomly allocated to receive: 1) usual care plus the patient decision aid or 2) usual care. For purposes of this study, usual care will include a booklet entitled, "Cystic fibrosis and lung transplantation" written by the Canadian Cystic Fibrosis Foundation plus any other written or educational material that the local CF centre normally provides.

ELIGIBILITY:
Inclusion Criteria:

* FEV less than or equal to 40% predicted

Exclusion Criteria:

* Patients unable to provide informed consent
* Patients on a lung transplant waiting list
* Patients who are lung transplant recipients
* Patients deemed too sick for transplant
* Only one sibling per family to minimize contamination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-09; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Knowledge, realistic expectations and decisional conflict 3 weeks after using the decision aid.

SECONDARY OUTCOMES:
Durability of the decision one year after the patient decision aid.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Aaron, MD FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Vandemheen KL, O'Connor A, Bell SC, Freitag A, Bye P, Jeanneret A, Berthiaume Y, Brown N, Wilcox P, Ryan G, Brager N, Rabin H, Morrison N, Gibson P, Jackson M, Paterson N, Middleton P, Aaron SD. Randomized trial of a decision aid for patients with cystic fibrosis considering lung transplantation. Am J Respir Crit Care Med. 2009 Oct 15;180(8):761-8. doi: 10.1164/rccm.200903-0421OC. Epub 2009 Jul 9. PMID 19590021